CLINICAL TRIAL: NCT01095614
Title: Impact of Women Hormonal Status (Oral Contraception vs no Contraception) on Substrate Utilization During Exercise
Brief Title: Substrate Utilization and Hormonal Status in Women
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: French Federation of Physical Education and Gymnastic (EPGV) (Unknown)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Other Study IDs: CHU-0068; AU818 (Other: CPP)
Record Dates: First submitted 2010-02-16; First posted 2010-03-30 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Substrate Utilization
Keywords: Women; Hormonal status; Exercise; Substrate utilization; Women Hormonal Status (with oral contraception or without any contraception)
MeSH Terms: conditions — Motor Activity

GROUPS / COHORTS (2):
- 12 women with oral contraception
- 12 women without any contraception

SUMMARY:
Women sexual hormones (i.e. estrogen) are involved in the regulation of substrate utilization and storage. Being under oral contraception (OC) may conduct to metabolic and hormonal modifications, but results are confused regarding the impact on substrate utilization. In the present study, the aim is then to explore the effect of hormonal status on substrate utilization during sous-maximal exercise, comparing women with and without OC.

We hypothesised that women under OC have a lower Respiratory Exchange Ratio (RER) at exercise than women without contraception underlying a greater reliance on fat oxidation.

DETAILED DESCRIPTION:
24 healthy young women (12 with OC and 12 without any contraception) will complete a maximal test on an ergometer cycle to obtain their maximal oxygen consumption (VO2max).Their body composition will be assessed by DXA. They will be asked to complete 3 experimental sessions.

During a first session the volunteers will remain inactive, and only a breakfast will be offered. During the second session, a breakfast will be offered and they will have to complete a sub-maximal exercise set at 60% of their VO2max 3 hours after breakfast. And the third session will consist in the realisation of exercise on fast state. Those three sessions will be realized in a randomized order. Several blood (catheter) and salivary samples will be collected during the three sessions, throughout the experimental day.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Adults between 19 to 30 years old
* Body mass index between 20 and 25 kg.m-²
* Oral contraception (half of the sample) : mini-dosed, and mono-phasic, ethinyl estradiol ≤ 30 µg
* Without contraception (half of the sample)
* Affiliated to National Health Insurance
* Subject giving her written informed consent
* Subject considered as normal after clinical examination and medical questionnaire.

Exclusion Criteria:

* Chronic pathologies : cardiovascular diseases, cancer, chronic inflammation diseases, renal, intestinal impairments
* Refusal to be registered on the National Volunteers Data file
* Being in exclusion on the National Volunteers Data file
* Practising intensive physical exercise
* Heavy consumer of alcohol or/and tobacco
* Previous medical and/or surgery judged by the investigator as incompatible with this study
* Pregnancy

Ages: 19 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 24 healthy young women (12 with OC and 12 without any contraception) will complete a maximal test on an ergometer cycle to obtain their maximal oxygen consumption (VO2max).Their body composition will be assessed by DXA. They will be asked to complete 3 experimental sessions
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Substrate utilization will be the main outcome under study.For each volunteer, it will be assessed during exercise (between 12h and 12h45) for the 2 experimental conditions with exercise | during exercise (between 12h and 12h45)
  Substrate utilization:
  The Respiratory Exchange Ratio (RER) that corresponds to carbon dioxide production divided by oxygen consumption (VCO2/VO2) will be used to determine the energetic substrate used during exercise. This RER will be obtained, in continuous, thanks to an indirect calorimetric system composed of a breath by breath gas analyzer. A RER closed to 0.7 illustrates lipid utilization while carbohydrate use will correspond to a RER that reached 1.

SECONDARY OUTCOMES:
The hormonal regulation involved in substrate utilization. It will be assessed during the 3 experimental conditions during all the experimental day: - Breakfast + exercise - Exercise alone - Breakfast alone | before (8h, 8h45), during (12h, 12h20, 12h30, 12h45) and after exercise (13h15, 13h45; 14h45)
  The hormonal regulations involved in the substrate utilization will be assessed thanks to blood samples collected before, during and after exercise.
  At each blood collection, the nurses will collect a EDTA tube (5ml) used to assess free fatty acid and glycerol; and 2 heparin ones (2*5ml) to assess 17β-œstradiol, progesterone, triglycerides, cholesterol, HDL-C, LDL-C, glucose, insulin, growth hormone, IGF-I, IGFBP-1, IGFBP-3, adrenaline, noradrenaline, Atrial Natriuretic Peptide, and C-Reactive Protein.

CONTACTS AND LOCATIONS:
Overall Officials: Martine DUCLOS, Pr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France